CLINICAL TRIAL: NCT01092104
Title: A Proof of Concept, Multiple Dose-Escalating Study to Evaluate the Antiviral Activity, Safety, and Pharmacokinetics of the CCR5 Antagonist TBR 652 in HIV 1-Infected, Antiretroviral Treatment-Experienced, CCR5 Antagonist-Naïve Patients
Brief Title: A Proof of Concept Study to Evaluate the Antiviral Activity, Safety, and Pharmacokinetics of the CCR5 Antagonist TBR 652 in HIV 1-Infected, Antiretroviral Treatment-Experienced, CCR5 Antagonist-Naïve Patients
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Tobira Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 652-2-201
Record Dates: First submitted 2010-03-22; First posted 2010-03-24 (Estimated); Last update posted 2013-07-10 (Estimated); Status verified 2013-07

CONDITIONS: HIV-1 Infection
MeSH Terms: interventions — cenicriviroc

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- TBR-652 25 mg QD (Experimental): TBR 25 mg QD for 10 days
  Interventions: Drug: TBR-652
- Placebo (Placebo Comparator): Matching Placebo QD for 10 days
  Interventions: Drug: TBR-652 Matching Placebo
- TBR-652 50 mg QD (Experimental): TBR-652 50 mg QD for 10 days
  Interventions: Drug: TBR-652 50 mg
- TBR-652 75 mg QD (Experimental): TBR-652 75 mg QD for 10 days
  Interventions: Drug: TBR-652 75 mg
- TBR-652 100 mg QD (Experimental): TBR-652 100 mg QD for 10 days
  Interventions: Drug: TBR-652 100 mg
- TBR-652 150 mg (Experimental): TBR-652 150 mg QD for 10 days
  Interventions: Drug: TBR-652 150 mg

INTERVENTIONS:
Drug: TBR-652 — TBR-652 25 mg
  Arms: TBR-652 25 mg QD
Drug: TBR-652 Matching Placebo — Matching Placebo
  Arms: Placebo
Drug: TBR-652 50 mg — TBR-652 50 mg QD for 10 days
  Arms: TBR-652 50 mg QD
Drug: TBR-652 75 mg — TBR-652 75 mg QD for 10 days
  Arms: TBR-652 75 mg QD
Drug: TBR-652 100 mg — TBR-652 100 mg QD for 10 days
  Arms: TBR-652 100 mg QD
Drug: TBR-652 150 mg — TBR-652 150 mg QD for 10 days
  Arms: TBR-652 150 mg

SUMMARY:
A double-blind, randomized, placebo-controlled, dose-escalating study to assess the antiviral activity, safety, tolerability, and pharmacokinetics (PK) of the CCR5 antagonist TBR 652 monotherapy dosed orally once daily (QD) for 10 days in HIV 1-infected, antiretroviral treatment-experienced, CCR5 antagonist-naïve patients.

ELIGIBILITY:
Inclusion Criteria:

1. No clinically significant findings on Screening evaluations (clinical, laboratory, and ECG), which in the opinion of the Investigator would interfere with the subject's ability to comply with the protocol.
2. Antiretroviral treatment-experienced; no antiretroviral therapy for at least 6 weeks prior to study entry.
3. CCR5 antagonist therapy naive.
4. CD4 cell count >/= 250 cells/mm3 during Screening (within 30 days prior to first dose).
5. Two separate qualifying plasma HIV 1 RNA levels >/= 5,000 copies/mL within 45 days prior to first dose.
6. Females who are not of reproductive potential (documented to be surgically sterile or postmenopausal [defined as amenorrhea ≥ 1 year and follicle stimulating hormone {FSH} ≥ 30 mU/mL]).
7. Females of child-bearing potential may be enrolled following a negative serum pregnancy test. If participating in activity that could lead to pregnancy, males and females shall agree to use two forms of barrier method contraception during the trial and for 2 months after stopping the medication.

Exclusion Criteria:

1. Presence of CXCR4- or dual/mixed-tropic HIV 1 virus.
2. Active CDC category C disease (except cutaneous Kaposi's sarcoma not requiring systemic therapy during the trial).
3. History of infection with hepatitis B or hepatitis C virus, history of cirrhosis, or any known active or chronic liver disease. NOTE: Hepatitis B vaccinated patients are eligible.
4. Serum ALT or AST values greater than Grade 1 or bilirubin values greater than the upper limit of normal (ULN) at Screening.
5. History of HIV-2.
6. Recent history (< 30 days prior to study drug administration) of clinically significant infection.
7. Pregnant females or females who are breastfeeding.
8. Treatment with immunomodulating agents (such as systemic corticosteroids, interleukins, interferons) or any agent with known anti-HIV activity within 30 days prior to study drug administration.
9. Treatment with any vaccine within 30 days of study drug administration.
10. A positive pre-study drug screen, including amphetamines, barbiturates, cocaine, or PCP.
11. Anticipated use of antacids during the trial and/or within 7 days prior to first dose of study drug.
12. Current alcohol or drug use, which in the expert judgment of the investigator, will interfere with the patient's ability to comply with the protocol requirements.
13. Inability, in the opinion of the investigator, to comply with the dosing schedule and protocol evaluations.
14. Use of any experimental medications within 4 weeks prior to Screening.
15. Current (within 30 days prior to the first dose of study drug) or anticipated use of antimetabolites; alkylating agents; or drugs, herbal preparations, and foods (including grapefruit) known to affect the CYP 3A4 or CYP 2C8 enzymes or P-glycoprotein transporters.
16. History of clinically significant hepatic, metabolic, endocrine, renal, hematologic, pulmonary, gastrointestinal, or cardiovascular disorders (including ECG abnormalities).
17. Uncontrolled hypertension.
18. Presence of a malabsorption syndrome affecting drug absorption (e.g., Crohn's disease, chronic pancreatitis).
19. History of malignancy with exception of cured basal or squamous cell carcinoma of the skin.
20. Receipt of radiation or cytotoxic chemotherapeutic agents and not recovered from side effects prior to the first dose of study medication.
21. Subjects who have used any over-the-counter medications (including phytotherapeutic, herbal, or plant-derived preparations) within 14 days prior to the first dose of study medication, unless approved by the Investigator, or who have used St. John's wort within 21 days prior to the first dose of study drug. (St. John's wort is prohibited during the study.)
22. History or presence of an abnormal ECG.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2009-02; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
HIV-1 RNA Change from Baseline | 10 days

REFERENCES:
- [Result] Lalezari J, Gathe J, Brinson C, Thompson M, Cohen C, Dejesus E, Galindez J, Ernst JA, Martin DE, Palleja SM. Safety, efficacy, and pharmacokinetics of TBR-652, a CCR5/CCR2 antagonist, in HIV-1-infected, treatment-experienced, CCR5 antagonist-naive subjects. J Acquir Immune Defic Syndr. 2011 Jun 1;57(2):118-25. doi: 10.1097/QAI.0b013e318213c2c0. PMID 21317794
- [Result] Marier JF, Trinh M, Pheng LH, Palleja SM, Martin DE. Pharmacokinetics and pharmacodynamics of TBR-652, a novel CCR5 antagonist, in HIV-1-infected, antiretroviral treatment-experienced, CCR5 antagonist-naive patients. Antimicrob Agents Chemother. 2011 Jun;55(6):2768-74. doi: 10.1128/AAC.00713-10. Epub 2011 Apr 12. PMID 21486960